CLINICAL TRIAL: NCT04891588
Title: Evaluation of Glaucoma or Ocular Hypertension Patients With Pre-existing Ocular Surface Disease Switched From a Preserved Prostaglandin Analog - Timolol Fixed Combination to a Preservative - Free Latanoprost - Timolol Fixed Combination
Brief Title: Switching From the Preserved to the Preservative - Free Latanoprost - Timolol FC in Glaucoma Patients With OSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR ZAG 02/21 AG 8.1-21/18-2; DRKS00024581 (Registry Identifier: DRKS - German Clinical Trials Register)
Record Dates: First submitted 2021-04-28; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular surface disease; preservative; treatment; Prostaglandin/timolol fixed combination; tolerability
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Switching the preserved to preservative free prostaglandin analog-timolol FC (Experimental): To switch preserved prostaglandin analog- timolol FC (Fixapost 50 micrograms/ml + 5 mg/ml eye drops, solution in single-dose container) in the period of three months in patients with ocular hypertension and open angle glaucoma who exhibit ocular surface disease (OSD) signs and symptoms to an equally effective and safe preservative - free (PF) latanoprost - timolol FC in order to investigate whether that can result in alleviation or elimination of OSD and improvement of local tolerability.
  Interventions: Drug: Switching the preserved prostaglandin analog-timolol FC to Fixalpost (preservative free prostaglandin analog-timolol FC)

INTERVENTIONS:
Drug: Switching the preserved prostaglandin analog-timolol FC to Fixalpost (preservative free prostaglandin analog-timolol FC) — switching preserved prostaglandin analog- timolol FC (fixed combination) in the period of three months in patients with ocular hypertension and open angle glaucoma who exhibit ocular surface disease (OSD) signs and symptoms to an equally effective and safe preservative - free (PF) latanoprost - timolol FC (Fixalpost).
  form: preservative free latanoprost - timolol fix combination (50 micrograms/ml latanoprost + 5 mg/ml timolol), ocular solution dosage: once daily, at 8.00 p.m. duration: 3 months
  Other Names: Fixalpost ( T2347), 50 micrograms/ml latanoprost + 5 mg/ml timolol maleate eye drops, solution in single-dose container

SUMMARY:
Glaucoma is a group of chronic eye diseases that are characterized by a progressive optic nerve damage and consequent visual loss. In most cases, it is associated with elevated intraocular pressure. If glaucoma left untreated, complete blindness can occur. Prostaglandin analog- timolol FCs are common glaucoma therapy because these drugs have been shown to effectively lower intraocular pressure (IOP). It is also known that chronic use of preservatives in the drops leads to ocular surface disease (OSD) which can lead to low tolerability of prescribed drops and gaps in the dosing regimen.

The purpose of this study is to investigate whether drug preservative elimination results in reduction of OSD symptoms and signs as well as improvement of latanoprost-timolol FC local tolerability in the treatment of glaucoma and ocular hypertension.

In this trial, on each visit (V1, V2 and V3) following tests will be used: Snellen visual acuity, IOP measurement by Goldman applanation tonometry, OSD signs assessment on the slit lamp (corneal and conjunctival fluorescein surface staining, conjunctival hyperemia and tear film stability assessment using Tear Break- up Time test - TBUT). Visual Analog Scale (VAS) will be used for a subjective assessment of drug tolerability. The association of quality of life and dry eye symptoms in participants will be measured by the Ocular Surface Disease Index (OSDI) questionnaire.

DETAILED DESCRIPTION:
Glaucoma is a heterogeneous group of chronic ocular diseases characterized by a loss of the retinal nerve fiber layer and consequent damage to the optic nerve head. Increased intraocular pressure is considered a major risk factor for development of the disease. If glaucoma left untreated, visual field impairment and complete visual loss can occur. Due to the effective reduction of intraocular pressure, prostaglandin analog-timolol fixed combinations (FC) are considered to be a mainstay in glaucoma treatment. However, it is well known that long-term use of preservatives in glaucoma drops leads to ocular surface disease (OSD) which causes low tolerability and nonadherence with prescribed therapy.

The study is designed to determine whether switching from a preserved prostaglandin analog- timolol FC to an equally effective and safe preservative - free latanoprost - timolol FC can result in alleviation or elimination of OSD and improvement of local tolerability.

In this study, on each visit (V1, V2 and V3) following tests will be performed: Snellen visual acuity, IOP measurement by Goldman applanation tonometry, OSD signs assessment on the slit lamp (fluorescein corneal and conjunctival fluorescein surface staining, conjunctival hyperemia and tear film stability assessment using Tear Break- up Time test -TBUT). The subjective evaluation of drug tolerability will be quantified by Visual Analog Scale (VAS). The evaluation of the association of quality of life and dry eye symptoms in respondents will be examined with the Ocular Surface Disease Index (OSDI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients with open angle galucoma or ocular hypertension that had been controlled (stable IOP <19mmHg) by commercially available preserved PGA -timolol FC for at least 3 months
* Stable visual field (based on at least two reliable visual field tests performed within the last 12 months)
* Central corneal thickness within the range 500-580µm.
* mild to moderate hyperaemia based on MacMonnies (scores 1 and 2)

Exclusion Criteria:

* Best-corrected visual acuity (BCVA) 0,1 or lower
* Severe visual field defects (MD 12 dB or higher)
* Any intraocular surgery (other than filtration surgery performed at least 6 months before screening)
* Any ocular surface abnormality preventing accurate IOP measurement
* Acute ocular inflammation
* Contact lens wearers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-09-08 (Estimated); Study Completion 2021-12-08 (Estimated)

PRIMARY OUTCOMES:
Change of drug tolerability | through study completion, an average of 6 months
  In this study, the following test is carried out at every visit (V1, V 2 and V3) every month to determine the change of drug tolerability:
  The Visual Analog Scale is used to determine drug tolerability.
Change of symptoms of ocular surface disease | through study completion, an average of 6 months
  In this study, the following tests is carried out at every visit (V1, V 2 and V3) every month to determine the change of symptoms of ocular surface disease:
  The subjects' symptoms of ocular surface disease is assessed using a standardized questionnaire - Ocular Surface Disease Index - OSDI questionnaire.
Change of visual function | through study completion, an average of 6 months
  In this study, the following tests is carried out at every visit (V1, V 2 and V3) every month to evaluate change of visual function:
  Visual Acuity Testing (Snellen Chart).
Change of signs of ocular surface disease | through study completion, an average of 6 months
  In this study, the following tests is carried out at every visit (V1, V 2 and V3) every month to determine the change of symptoms of ocular surface disease:
  Slit lamp examination (fluorescein staining of the cornea and conjunctiva, hyperemia of the conjunctiva)
Change of tear film stability | through study completion, an average of 6 months
  In this study, the following tests is carried out at every visit (V1, V 2 and V3) every month to evaluate change of signs of ocular surface disease:
  assessment of the tear film stability by measuring the tear film break-up time (TBUT).

SECONDARY OUTCOMES:
Evaluation of the effectiveness of preservative-free latanoprost / timolol FC in terms of changing intraocular pressure values | through study completion, an average of 6 months
  In this study, applanation tonometry according to Goldmann will be performed at every visit (V1, V 2 and V3) every month to measure intraocular pressure in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Jandroković, MD PhD, Principal Investigator — Klinički Bolnički Centar Zagreb
Locations (1):
- Klinički bolnički centar Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xing Y, Zhu L, Zhang K, Huang S. The efficacy of the fixed combination of latanoprost and timolol versus other fixed combinations for primary open-angle glaucoma and ocular hypertension: A systematic review and meta-analysis. PLoS One. 2020 Feb 27;15(2):e0229682. doi: 10.1371/journal.pone.0229682. eCollection 2020. PMID 32106236
- [Background] Uusitalo H, Chen E, Pfeiffer N, Brignole-Baudouin F, Kaarniranta K, Leino M, Puska P, Palmgren E, Hamacher T, Hofmann G, Petzold G, Richter U, Riedel T, Winter M, Ropo A. Switching from a preserved to a preservative-free prostaglandin preparation in topical glaucoma medication. Acta Ophthalmol. 2010 May;88(3):329-36. doi: 10.1111/j.1755-3768.2010.01907.x. PMID 20546237
- [Background] Misiuk-Hojlo M, Pomorska M, Mulak M, Rekas M, Wierzbowska J, Prost M, Wasyluk J, Lubinski W, Podboraczynska-Jodko K, Romaniuk W, Kinasz R, Ortyl-Markiewicz R, Mocko L, Zaleska-Zmijewska A, Rokicki D, Baudouin C. The RELIEF study: Tolerability and efficacy of preservative-free latanoprost in the treatment of glaucoma or ocular hypertension. Eur J Ophthalmol. 2019 Mar;29(2):210-215. doi: 10.1177/1120672118785280. Epub 2018 Jul 12. PMID 29998767
- [Background] Guven Yilmaz S, Degirmenci C, Karakoyun YE, Yusifov E, Ates H. The efficacy and safety of bimatoprost/timolol maleate, latanoprost/timolol maleate, and travoprost/timolol maleate fixed combinations on 24-h IOP. Int Ophthalmol. 2018 Aug;38(4):1425-1431. doi: 10.1007/s10792-017-0601-8. Epub 2017 Jun 14. PMID 28616797